CLINICAL TRIAL: NCT05903677
Title: The Relationship Between Preoperative Levels of Ionized Magnesium and Risk of Acute Kidney Injury After Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Ahmed Kaleed Abdelhalim, Resident doctor, Assiut University
Other Study IDs: Preoperative magnesium and AKI
Record Dates: First submitted 2023-06-02; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Magnesium Disorder
MeSH Terms: interventions — Blood Urea Nitrogen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults undergoing cardiac surgery without preoperative renal affection: Detect the preoperative magnesium levels in adults undergoing cardiac surgery without preoperative renal affection and follow up if they developed postoperative acute kidney injury or not.
  Interventions: Other: magnesium levels

INTERVENTIONS:
Other: magnesium levels — Detection of the relationship between cardiac surgery associated AKI and preoperative magnesium levels.
  Other Names: Serum creatinine and blood urea nitrogen (BUN)

SUMMARY:
Detection the relationship between preoperative ionized magnesium levels and the risk of acute kidney injury after cardiac surgery.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a major medical problem that is of particular concern after cardiac surgery. The reported prevalence of cardiac surgery-associated acute kidney injury (CSA-AKI) is up to 30% and is independently associated with an increase of morbidity and mortality .So this study is for measuring preoperative ionized magnesium levels of patients who will undergo cardiac surgeries then measuring postoperative serum creatinine, BUN and urine output to detect if they developed AKI or not and if there is a relationship between the post cardiac surgery AKI and preoperative ionized magnesium levels.

ELIGIBILITY:
Inclusion Criteria:

1. patients more than or equal 18 yrs.
2. patients undergoing cardiac surgery between July 2023 and July 2024

Exclusion Criteria:

1. patients with known Kidney disease.
2. patients less than 18 yrs

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: people more than or equal 18 years who undergo open heart surgery between July 2023 to July 2024 and not known to have kidney disease .
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Post cardiac surgery AKI according to KDIGO criteria with low preoperative magnesium level | Baseline
  Measuring preoperative magnesium level and postoperative kidney functions in form of serum creatinine in umol/L , BUN in mmol/L and urine output ml/h to detect the relationship between preoperative low magnesium level and risk of acute kidney injury after cardiac surgery.
Post cardiac surgery AKI according to KDIGO criteria with normal or high preoperative magnesium level | basline
  Measuring preoperative magnesium level and postoperative serum creatinine, BUN and urine output to detect the relationship between preoperative magnesium level and risk of acute kidney injury after cardiac surgery.
Post cardiac surgery normal kidney functions with low preoperative magnesium level | basline
  Measuring preoperative magnesium level and postoperative serum creatinine, BUN and urine output to detect the relationship between preoperative magnesium level and risk of acute kidney injury after cardiac surgery.

REFERENCES:
- [Background] Koh HB, Jung CY, Kim HW, Kwon JY, Kim NH, Kim HJ, Jhee JH, Han SH, Yoo TH, Kang SW, Park JT. Preoperative Ionized Magnesium Levels and Risk of Acute Kidney Injury After Cardiac Surgery. Am J Kidney Dis. 2022 Nov;80(5):629-637.e1. doi: 10.1053/j.ajkd.2022.03.004. Epub 2022 Apr 23. PMID 35469966